CLINICAL TRIAL: NCT06255457
Title: Mechanisms and Outcomes in Patients With Arrhythmic Mitral Valve Prolapse Undergoing Mitral Valve Surgery
Brief Title: Ventricular Arrhythmias in Patients Undergoing Mitral Valve Surgery
Acronym: Mitra-VT
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Bahira Shahim, Assistant professor, Karolinska Institutet
Other Study IDs: VR 2022-01472; SG-23-0142-B (Other Grant/Funding Number: Svenska Sällskapet för Medicinsk Forskning (SSMF)); 987010 (Other Grant/Funding Number: Svenska Läkaresällskapet (SLS)); 20220524 (Other Grant/Funding Number: Hjärtlungfonden (HLF)); 2-116/2023 (Other Grant/Funding Number: karolinska Institutet)
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mitral Regurgitation; Mitral Valve Prolapse; Ventricular Tachycardia
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Arrhythmogenic mitral valve prolapse versus non-arrhythmogenic mitral valve prolapse: Surgical repair or replacement of the mitral valve due to significant mitral regurgitation according to standard of care.
  Interventions: Procedure: Mitral valve surgery

INTERVENTIONS:
Procedure: Mitral valve surgery — Mitral valve repair or replacement of mitral regurgitation

SUMMARY:
Study objectives:

* To assess the impact of mitral valve surgery for mitral regurgitation on ventricular arrhythmic burden and surrogate markers of fibrosis in patients with arrhytmogenic mitral valve prolapse (MVP) from baseline to 6 months after surgery
* To characterize the molecular landscape of arrhytmogenic MVP

Study design:

-Prospective explorative observational study

Study population:

-90 patients with arrhytmogenic MVP and without arrhytmogenic MVP (controls) eligible for mitral valve surgery for mitral regurgitation will be enrolled. All patients will be evaluated with cardiac magnetic resonance (CMR) imaging and continuous seven day arrhythmic monitoring before and at 6 months after mitral valve surgery

DETAILED DESCRIPTION:
Prospective explorative observational study in which the impact of mitral valve surgery for mitral regurgitation on ventricular arrhytmias and CMR imaging biomarkers will be examined in patients with arrhythmogenic MVP compared to those without arrhythmogenic MVP (controls). Molecular phenotyping of endocardial biopsies in patients with and without arrhythmogenic MVP will be performed as well as molecular phenotyping of the myxomatous disease in explanted valves by means of deep RNA single cell sequencing. Using CMR in 90 patients with MVP before and 6 months after mitral valve surgery, the presence and type (reversible vs irreversible) of papillary muscle and cardiac fibrosis will be characterized. To assess change in ventricular arrhytmic burden after surgery, patients will undergo continuous seven day monitoring with E-patch at baseline and at 6 months after mitral valve surgery. During surgery, explanted mitral valves (in patients undergoing replacement) as well as endocardial biopsies will be collected.

ELIGIBILITY:
Inclusion criteria

* Age 18 and over
* Patients with and without (controls) arrhythmogenic MVP in need of mitral valve surgery for primary mitral regurgitation according to current standard of care

Exclusion criteria

* Secondary mitral regurgitation
* Primary mitral regurgitation not due to degenerative disease (including rheumatic disease)
* Co-existing moderate or severe aortic valve disease
* Congenital heart disease
* Inherited or acquired cardiomyopathy
* Non-incidental or symptomatic coronary artery disease
* Uncontrolled atrial fibrillation (resting heart rate > 100/min)
* Pregnancy
* Unable to undergo CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with and without arrhythmogenic MVP with primary mitral regurgitation eligible for mitral valve surgery according to current standard of care.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular arrhythmias | 6 months
  Change in ventricular arrhythmic burden (composite of non-sustained or sustained ventricular tachycardias, ventricular fibrillation or premature ventricular complexes)
Extracellular volume | 6 months
  Change in indexed extracellular volume as surrogate marker for diffuse reversible fibrosis measured by CMR

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Univeristy Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No